CLINICAL TRIAL: NCT07047677
Title: Ex Vivo Evaluation of Experimental Radiolabeled Ligand Binding in Human Tissue Using Autohistoradiography HERO (Human Ex-vivo RadiOligand) Platform
Brief Title: Ex Vivo Evaluation on Human Tissue of the Binding of Experimental Radiolabeled Ligands
Acronym: HERO
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2025PI088
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Tissue Model

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Early assessment of tissue uptake of experimental ligands — Ex vivo evaluation of the binding of experimental radiolabeled ligands on human tissue using autohistoradiography

SUMMARY:
The HERO project aims to structure an ex vivo screening platform, based on anonymized human tissues, to early assess the tissue fixation of experimental ligands in an ethical, translational approach that complies with the principles of the 3Rs (Replacement, Reduction, Refinement).

DETAILED DESCRIPTION:
The development of radioligands targeting structures of diagnostic or therapeutic interest is a central challenge in nuclear medicine. However, their selection still relies primarily on animal models, which are poorly representative of human tissue, limiting clinical transposability and delaying innovation, in contradiction with the ethical principles of animal experimentation.

Recent work has highlighted the value of ex vivo approaches on human tissue to better anticipate the specificity of radioligand binding, while reducing the need for animal models. Autohistoradiography, in particular, allows precise visualization of the tissue distribution of radiolabeled molecules, without systemic interference.

The HERO project aims to structure an ex vivo screening platform, based on anonymized human tissues, to early assess the tissue fixation of experimental ligands in an ethical, translational approach that complies with the principles of the 3Rs (Replacement, Reduction, Refinement).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgical resection at the Nancy University Hospital after 2019 (Information provided in the welcome booklet or on posters displayed in waiting rooms, mentioning the possible use of data or resection specimens, unless otherwise stated).
* No documented objection, in accordance with the MR004 methodology.
* Frozen human tissues (slides, blocks, or sections) from surgical resection or biopsy, transmitted by the CRB or the biopathology department.
* Samples are fully anonymized before being made available for analysis.

Exclusion Criteria:

* • Unusable tissue (degraded, insufficient, contaminated, poorly preserved).

  * Lack of traceability of the material.
  * Explicit opposition from the patient to the use of their tissue for research.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum of 300 human tissue samples will be analyzed over a period of 5 years.
  This volume allows for the exploration of a variety of tissue types (tumor, inflammatory, healthy) and the testing of several types of radiolabeled molecules, while ensuring adequate reproducibility for each experimental condition.
  The samples will be provided by the Pathology Department of the Nancy University Hospital, in compliance with regulatory and ethical procedures.
  Each sample will undergo one or more ex vivo autohistoradiography analyses, without the need for any new samples.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Ex vivo evaluation of the binding of experimental radiolabeled ligands on human tissue by autohistoradiography | 10 days
  Signal /background noise ration, in region of interest

SECONDARY OUTCOMES:
Identify specific tissue fixation profiles according to the nature of the molecules (Antibodies, peptides, nanobodies, etc.). | 1 day
  Signal/background noise ratio (calculated between the target area and a healthy area on the same slice).
Compare the biodistribution of the molecule of interest between different types of tissues (tumor, inflammatory, healthy, etc.). | 10 days
  Analysis of biodistribution across the entire section (depending on the nature of the tissue).
Identify ligands exhibiting specific and relevant tissue binding, warranting further in vivo evaluation. | 1 year
  Inter-tissue differences (tumor, inflammatory, healthy tissue, etc.) for the same molecule.